CLINICAL TRIAL: NCT06311994
Title: Applicability and Efficiency of Virtual Reality Intervention in Knee Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Aydanur Aydin, Assist.Prof.Dr., Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GumushaneUni
Record Dates: First submitted 2024-02-17; First posted 2024-03-15 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-03

CONDITIONS: Virtual Reality; Symptom Management; Surgery; Quality of Life

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with virtual reality (Experimental): Factors that may affect patient compliance with the "VR-based intervention" method to be applied to patients undergoing knee surgery and the factors that may affect the measurements were evaluated through a literature review and inclusion and exclusion criteria were created.
  Interventions: Device: Virtual reality
- Control (No Intervention): Among the randomized patients, patients included in the control group will be included in the conventional rehabilitation program.

INTERVENTIONS:
Device: Virtual reality — Factors that may affect patient compliance with the "VR-based intervention" method to be applied to patients undergoing knee surgery and the factors that may affect the measurements to be performed were evaluated through a literature review and inclusion and exclusion criteria were created.
  Arms: Intervention with virtual reality

SUMMARY:
The stress experienced by patients in hospital environments can lead to a range of issues, from clinical decision-making to discharge. Although stress levels can contribute to new problems, individual characteristics also play a significant role in clinical recovery. Knee surgery is a commonly performed procedure in our country that provides patients with an effective solution to joint-related issues. However, stress experienced by patients who undergo surgery can have negative consequences, from managing problems during their hospital stay to their overall quality of life. The search for effective stress management methods is ongoing and has gained momentum with the development of new technological products. Virtual reality (VR) applications are a novel approach in the literature for managing various issues. Research is being conducted in different areas of our country using this approach. The aim of this project is to evaluate the feasibility, acceptability, and effectiveness of different environment perceptions using virtual reality glasses on postoperative mobilization and well-being in individuals undergoing knee surgery for the first time. The project sample is a randomized controlled trial consisting of 30 patients who will undergo orthopedic surgery for the first time at the Gümüşhane State Hospital orthopedic clinic and meet the acceptance criteria. In the intervention group, patients will view relaxing virtual environment images with VR glasses after surgery. Following the relaxation session, participants will be presented with content to exercise in the virtual environment. Patients will be instructed to perform breathing exercises set in forest and underwater scenes to aid relaxation. The effectiveness of the intervention will be assessed using the Tampa Kinesiophobia Scale and Patient Mobility Scale. A satisfaction scale with a linear format will be used to evaluate the acceptability of the intervention. In addition, a data collection form, developed by the researcher, will be used to gather information on participant characteristics. The obtained data will be analyzed using t-tests, analysis of variance, correlation, and regression tests. Currently, there is a growing number of studies that explore the relationship between technology and health. This project aims to investigate the impact of virtual reality glasses on symptom management. If the results are positive, this method could be used as a solution for various situations where individuals experience symptoms. The goal is to develop a usable product for postoperative mobilization based on the research findings.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being 18 years or older,
* This is the first time he's had knee surgery.

Exclusion Criteria:

* Not having a condition that prevents them from communicating, answering the questions asked in the research and participating in measurements,
* Having a physical problem that prevents arm movement (amputation, joint restriction in the extremities, etc.),
* Not having a chronic pain problem,
* Having hearing-vision problems,
* Having migraine, vertigo and active nausea problems,
* Do not have any problems (head wound, etc.) that would prevent the VR headset,
* Do not have claustrophobia,
* Being under psychiatric treatment,
* There is no history of epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain measure | 1 year
  VAS
Stress | 1 year
  Distress termometer

SECONDARY OUTCOMES:
Mobilization | 1 year
  Tampa Kinesiophobia Scale
Mobility | 1 year
  Patient Mobility Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Goh GS, Lohre R, Parvizi J, Goel DP. Virtual and augmented reality for surgical training and simulation in knee arthroplasty. Arch Orthop Trauma Surg. 2021 Dec;141(12):2303-2312. doi: 10.1007/s00402-021-04037-1. Epub 2021 Jul 15. PMID 34264380
- [Result] Leon-Munoz VJ, Moya-Angeler J, Lopez-Lopez M, Lison-Almagro AJ, Martinez-Martinez F, Santonja-Medina F. Integration of Square Fiducial Markers in Patient-Specific Instrumentation and Their Applicability in Knee Surgery. J Pers Med. 2023 Apr 25;13(5):727. doi: 10.3390/jpm13050727. PMID 37240897